CLINICAL TRIAL: NCT06046521
Title: A Clinical Study on the Effects of Temporomandibular Joint Dysfunction-Induced Limitations in Mouth Opening on Objective and Subjective Vocal Measurements
Brief Title: Impact of Temporomandibular Joint Dysfunction on Objective and Subjective Vocal Measures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ferit Bayram, Principal Investigator, Marmara University
Other Study IDs: MUDHF_PTT_03
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Temporomandibular Joint Disorders; Voice Change
MeSH Terms: conditions — Temporomandibular Joint Disorders; Dysphonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study aims to investigate the impact of temporomandibular joint dysfunction (TMD) on objective and subjective vocal parameters and the quality of life in affected patients. TMD is a pervasive public health issue that impacts approximately 25% of the general population and is notably more prevalent among women. The etiology of TMD is multi-factorial, with known risk factors such as parafunctional habits, emotional stress, occlusion issues, and orthodontic treatments. Internal derangements of the temporomandibular joint are the most common subtype of TMD, characterized by symptoms such as pain, joint noises, restricted mouth opening, and masticatory dysfunction.

This study particularly focuses on the limitations in mouth opening due to TMD and its effects on vocal characteristics and quality of life. Conservative treatment methods, such as non-steroidal anti-inflammatory drugs (NSAIDs) and occlusal splints, have been effective in symptom management unless there is clear evidence of joint collapse or ankylosis. The null hypothesis (H0) posits that the restriction in mouth opening has no impact on vocal parameters or quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 65 years.
* Capable of giving informed consent.
* Fluent in the local language for effective communication.
* No history of hearing impairment or high communicative demands in their profession.
* Absence of a history of vocal disorders or conditions affecting voice quality.

Exclusion Criteria:

* Individuals with a vocal disorder.
* Unable to provide informed consent or meet study requirements.
* Pregnant or lactating women.
* Presence of any medical condition that could potentially affect voice quality.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population comprises individuals aged between 18 and 65 who are fluent in the local language and capable of giving informed consent. Participants are screened to ensure they do not have a history of hearing impairment or high communicative demands in their profession. Moreover, individuals with a history of vocal disorders or any conditions that may affect voice quality are excluded from the study. The population also excludes pregnant or lactating women and individuals who are unable to provide informed consent or meet the study's specific requirements.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-04-14 (Estimated); Study Completion 2024-06-14 (Estimated)

PRIMARY OUTCOMES:
Change in Acoustic Voice Analyze measurements (Analysis of dysphonia in speech and voice) | T0: before occlusal splint treatment, T1: 1 month later occlusal splint treatment T2: 3 month later occlusal splint treatment T3: 6 months later occlusal splint treatment.
  Analysis of dysphonia in speech and voice (ADSV), asseses frequency domain parameters. It is based on 2 different vowels ((/a/ and /i/) from Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V) and 6 different sentences. Each sentence includes a separate voice analysis, such as whether it has all the vowels, if it makes glottal attack sounds or not, nasal sounds or explosive sounds.
Change in Acoustic Voice Analyze measurements (Motor Speech Profile) | T0: before occlusal splint treatment, T1: 1 month later occlusal splint treatment T2: 3 month later occlusal splint treatment T3: 6 months later occlusal splint treatment.
  Motor Speech Profile (MSP), is utilized to ensure that speech is produced with accuracy and precision. Oral-diadochokinetic performance that is unreliable, inconsistent, or aberrant may be a sign of problems with the central nervous system or with peripheral sensory-motor processes. The software is built on a variety of protocols that offer various motor speech patterns, including oral diadochokinetic (DDK) rate, second formant transition rate, and syllable rate.
Change in Acoustic Voice Analyze measurements (Acoustic Voice Quality Index) | T0: before occlusal splint treatment, T1: 1 month later occlusal splint treatment T2: 3 month later occlusal splint treatment T3: 6 months later occlusal splint treatment.
  Acoustic Voice Quality Index (AVQI, evaluates the voice signal's perceived quality. It is based on assessing a number of acoustic factors that are known to be connected to how well speech is received. These criteria include assessments of the signal's loudness, pitch, and spectral tilt as well as its level of noise and other aberrations.
Change in Acoustic Voice Analyze measurements (Acoustic Phonetic Analyzes) | T0: before occlusal splint treatment, T1: 1 month later occlusal splint treatment T2: 3 month later occlusal splint treatment T3: 6 months later occlusal splint treatment.
  Acoustic Phonetic Analyzes, voiced, non-voiced, bursting, fricative sounds are being consisted differently. Periodic glottal vibrations make a sound voiced. Non-voiced ones is produced with burs or frication. Voice on-set time measures glottal vibrations and periods. 12 words which include 4 vowels and 6 consonants will analyze via Praat. Spectrum analyzes of the fricative consonants will be done with spectral moments.
Change in Acoustic Voice Analyze measurements (Resonance Analyzes) | T0: before occlusal splint treatment, T1: 1 month later occlusal splint treatment T2: 3 month later occlusal splint treatment T3: 6 months later occlusal splint treatment.
  For the analyze the resonance disturbances, nasometer is being used and the scores calculate with a special formula which include nasal and oral acoustic energies. Oral, nasal and oro-nasal paragraphs will be used for production.

SECONDARY OUTCOMES:
Change in Oral Health Impact Profile-14 (OHIP-14): | T0: before occlusal splint treatment, T1: 1 month later occlusal splint treatment T2: 3 month later occlusal splint treatment T3: 6 months later occlusal splint treatment.
  Oral health related life quality is an individual's self perception of how his/her oral health influences his/her life quality. OHIP basically has 14 questions that can be categorized into scales as functional limitation, physical pain, psychological discomfort, physical, psychological and social insufficiency and handicap.
Influence of Clinical Case Report Changes (Painless unassisted mouth opening distance) | T0: before occlusal splint treatment, T1: 1 month later occlusal splint treatment T2: 3 month later occlusal splint treatment T3: 6 months later occlusal splint treatment.
  Painless unassisted mouth opening distance, patient will be asked open mouth freely and painless and then will be measured interincisal distance with using millimetric ruler and add overbite distance.
Influence of Clinical Case Report Changes (Maximum unassisted mouth opening distance) | T0: before occlusal splint treatment, T1: 1 month later occlusal splint treatment T2: 3 month later occlusal splint treatment T3: 6 months later occlusal splint treatment.
  Maximum unassisted mouth opening distance, patient will be asked to open mouth as much as possible. At that point, will questioned about feeling pain and if answer is yes where to feel. Muscle or junction, unilateral or bilateral pain situation will be saved. Finally overbite distance will be added.
Influence of Clinical Case Report Changes (Maximum assisted mouth opening distance) | T0: before occlusal splint treatment, T1: 1 month later occlusal splint treatment T2: 3 month later occlusal splint treatment T3: 6 months later occlusal splint treatment.
  Maximum assisted mouth opening distance, after completed maximum unassisted mouth opening, thumb will be placed on maxillary incisal teeth and index finger on mandibular incisal teeth and will try to open the patient's mouth and saved with adding overbite distance.
Influence of Clinical Case Report Changes (Vertical movement distances) | T0: before occlusal splint treatment, T1: 1 month later occlusal splint treatment T2: 3 month later occlusal splint treatment T3: 6 months later occlusal splint treatment.
  Vertical movement distances, at maximum intercuspal position, where the maxillary incisors cover the mandibular incisor is marked and distance to the incisal edge is saved as overbite. And at this position, distance between the maxillary and mandibulary incisors horizontally will be measured with the ruler and saved as overjet.
Influence of Clinical Case Report Changes (Way of movement) | T0: before occlusal splint treatment, T1: 1 month later occlusal splint treatment T2: 3 month later occlusal splint treatment T3: 6 months later occlusal splint treatment.
  Way of movement, patient will wait in a relax situation and open mouth as much as they can even if painful. While the mandible moves, observer will look at the deflection from the midline or at the last stage of opening deviation from the midline.
Influence of Clinical Case Report Changes (Eccentric movement distances) | T0: before occlusal splint treatment, T1: 1 month later occlusal splint treatment T2: 3 month later occlusal splint treatment T3: 6 months later occlusal splint treatment.
  Right and left lateral movement, while mouth slight open, at the maximum movement to the right side distance between the incisors will be measured with millimetric ruler and repeat the same movement for the left side.
Influence of Clinical Case Report Changes (Right and left movement) | T0: before occlusal splint treatment, T1: 1 month later occlusal splint treatment T2: 3 month later occlusal splint treatment T3: 6 months later occlusal splint treatment.
  Right and left lateral movement, while mouth slight open, at the maximum movement to the right side distance between the incisors will be measured with millimetric ruler and repeat the same movement for the left side.
Influence of Clinical Case Report Changes (Protrusion) | T0: before occlusal splint treatment, T1: 1 month later occlusal splint treatment T2: 3 month later occlusal splint treatment T3: 6 months later occlusal splint treatment.
  Protrusion, patient will be asked the open mouth slightly but wide enough to avoid inflict between incisors and move the mandible forward as much as possible. Space between the incisors will be measured.
Influence of Clinical Case Report Changes (Midline deviation) | T0: before occlusal splint treatment, T1: 1 month later occlusal splint treatment T2: 3 month later occlusal splint treatment T3: 6 months later occlusal splint treatment.
  Midline deviation, if the distance between the midline projections of the lower and upper jaws is more than 1 mm, the amount will be recorded along with the direction of shift.
Influence of Clinical Case Report Changes (Sounds of articulate) | T0: before occlusal splint treatment, T1: 1 month later occlusal splint treatment T2: 3 month later occlusal splint treatment T3: 6 months later occlusal splint treatment.
  Sounds of articulate, palpation bilaterally on the preauricular region will be done with two index finger and look at if there is a sound while patient opens and closes the mouth. If there is, what kind of sound is being heard will be specified between click, hard crepitation, soft crepitation, and no sound.
Influence of Clinical Case Report Changes (Pain scores after palpations of the TMJ and muscles of mastication) | T0: before occlusal splint treatment, T1: 1 month later occlusal splint treatment T2: 3 month later occlusal splint treatment T3: 6 months later occlusal splint treatment.
  Pain scores after palpations of the TMJ and muscles of mastication, palpation of muscles will be done while mouth is rest, there is a space between teeth and muscles are passive. Patient will be asked to feel any pain during palpation and score to mild, moderate, severe or none. And palpation of TMJ will be done through ear way and lateral side while patient opens and closes the mouth.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided